CLINICAL TRIAL: NCT01440972
Title: Assessment of Efficacy of Low Intensity Resistance Training in Women at Risk for Symptomatic Knee Osteoarthritis
Acronym: PBFR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: The American Geriatrics Society (Other)
Responsible Party: Principal Investigator, Neil A Segal, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 201109738
Record Dates: First submitted 2011-09-21; First posted 2011-09-27 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-10

CONDITIONS: Knee Osteoarthritis; Symptomatic Knee Osteoarthritis
Keywords: knee osteoarthritis; symptomatic knee osteoarthritis; isotonic leg-press strength; isokinetic knee extensor strength; quadriceps volume
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise without PBFR (Active Comparator)
  Interventions: Other: low intensity resistance training
- exercise with PBFR (Experimental)
  Interventions: Other: partial blood flow restriction (PBFR)

INTERVENTIONS:
Other: partial blood flow restriction (PBFR) — low intensity resistance training with partial blood flow restriction 3 times/week for 4 weeks.
  Arms: exercise with PBFR
Other: low intensity resistance training — low intensity resistance training without partial blood flow restriction
  Arms: Exercise without PBFR

SUMMARY:
The purpose of this study is to asses the efficacy of a 4 week low-intensity resistance training program with concurrent application of partial blood flow restriction (PBFR) to the exercising limbs to improve quadriceps strength and size, leg muscle power, and mobility in women at risk for developing symptomatic knee osteoarthritis. The primary outcome will be change in isotonic double leg-press 1 repetition maximum (1RM) strength. The investigators will test the following hypotheses. In comparison with low-intensity resistance training without use of PBFR, a four-week low-intensity resistance-training program with PBFR will:

Primary Hypothesis: Increase (a) double leg-press 1RM strength and (b) isokinetic knee extensor strength

Secondary Hypotheses:

1. Increase quadriceps muscle volume assessed by MRI
2. Increase lower limb muscle power on (a) double leg-press at 40% 1RM and (b) a timed stair climb
3. Not adversely effect knee pain or quality of life assessed by the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 45-65
* BMI greater than or equal to 25 kg/m2, or a history of a knee joint injury or surgery, or knee symptoms (pain, aching, or stiffness) on most of the last 30 days, or knee osteoarthritis

Exclusion Criteria:

* Resistance training at any time in the last 3 months prior to study
* Bilateral knee replacement
* Lower limb amputation
* Lower limb surgery in the last 6 months that affects walking ability or ability to exercise
* Back, hip or knee problems that affect walking ability or ability to exercise
* Unable to walk without a cane or walker
* Inflammatory joint or muscle disease such as rheumatoid or psoriatic arthritis or polymyalgia rheumatica
* Multiple sclerosis
* Known neuropathy
* Self-report of Diabetes
* Currently being treated for cancer or having untreated cancer
* Terminal illness (cannot be cured or adequately treated and there is a reasonable expectation of death in the near future)
* Peripheral Vascular Disease
* History of myocardial infarction or stroke in the last year
* History of deep venous thrombosis
* Chest pain during exercise or at rest
* Use of supplemental oxygen
* Inability to follow protocol (e.g. lack of ability to attend visits or understand instructions)
* Staff concern for subject health (such as history of dizziness/faintness or current restrictions on activity)
* Concurrent study participation (such as the MOST study)
* Unable to attend more than 2 days within any 1 week or unable to attend 4 or more sessions during the study

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Without PBFR | Exercise With PBFR
Started | 24 | 21
Completed | 21 | 19
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Without PBFR | Exercise With PBFR | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (6.9) | 56.1 (5.9) | 55.4 (6.5)
Gender [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Isotonic Double Leg-press 1 Repetition Maximum Strength Scaled to Body Mass
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: kg per kg body mass
Arm/Group | Exercise Without PBFR | Exercise With PBFR
Number analyzed (Participants) | 21 | 19
kg per kg body mass | 0.2 (0.3) | 0.4 (0.3)

2. Secondary Outcome: Change in Quadriceps Muscle Volume by Magnetic Resonance Imaging
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Exercise Without PBFR | Exercise With PBFR
Number analyzed (Participants) | 21 | 19
Percent change | 0.01 (.73) | 1.3 (0.80)

3. Secondary Outcome: Change in Lower Limb Muscle Power by Double Leg-press at 40% 1 Repetition Maximum
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Exercise Without PBFR | Exercise With PBFR
Number analyzed (Participants) | 21 | 19
Watts | 0.42 (.26) | .62 (.27)

4. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome Score Pain Subscale
Description: KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life QOL. The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. KOOS is patient-administered, the format is user friendly, and takes about 10 minutes to fill out. Only the pain sub scale was used for the reported study.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Without PBFR | Exercise With PBFR
Number analyzed (Participants) | 21 | 19
units on a scale | 1.8 (2.7) | 2.0 (2.8)

5. Secondary Outcome: Change in Isokinetic Knee Extensor Strength
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: Nm/kg
Arm/Group | Exercise Without PBFR | Exercise With PBFR
Number analyzed (Participants) | 21 | 19
Nm/kg | -0.05 (0.03) | .07 (.03)

ADVERSE EVENTS:
Arm/Group | Exercise Without PBFR | Exercise With PBFR
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No